CLINICAL TRIAL: NCT03022630
Title: The Creation of Models for Palliative Assessments to Support Severe Illness (COMPASS) Investigation: Testing Early and Ongoing Implementation of Palliative Care for Incurable Non-malignant Diseases
Brief Title: Palliative Care for Non-Malignant Diseases (COMPASS Trial)
Acronym: COMPASS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Gordon Bernard, Study Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 160746
Record Dates: First submitted 2016-06-03; First posted 2017-01-16 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-08

CONDITIONS: Liver Diseases; Liver Cirrhosis; NASH (Non-Alcoholic Steatohepatitis)
Keywords: palliative care; cirrhosis; liver disease; hepatology; end of life care; supportive care
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis; Non-alcoholic Fatty Liver Disease; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Palliative Care services (Other): Comprehensive Palliative Care services in addition to usual hepatic care
  Interventions: Other: Comprehensive Palliative Care services
- Usual hepatic care (Other): Usual hepatic care
  Interventions: Other: Usual hepatic care

INTERVENTIONS:
Other: Comprehensive Palliative Care services — Participants who are randomly assigned to the intervention arm will receive informational materials, comprehensive inpatient palliative care consultations with a palliative care physician or nurse practitioner, in addition to standard hepatic care. If the patient is discharged, follow-up consults will be provided by a palliative care nurse via telephone contact. Telephone contacts will occur on a flexible schedule (e.g., weekly, bi-weekly, monthly) based on the needs and wishes of the patient, at a minimum frequency of once a month. If a need for further care is identified from a telephone contact, appropriate follow-up (referral, appointment, clinical communication, etc.) will occur per standard procedures. If the participant is readmitted, the consultation schedule will restart.
  Arms: Comprehensive Palliative Care services
Other: Usual hepatic care — Participants randomized to the usual care arm will not be scheduled to meet with the palliative care service unless a consult is requested by the patient, the family, or treating physician. These consultations would include the same palliative care services as the intervention arm, excluding the informational patient materials and telephone consultations.
  Arms: Usual hepatic care

SUMMARY:
The purpose of this study is to evaluate, through a randomized controlled trial, the impact of integrated comprehensive palliative care services on time to first hospital readmission and other hospital utilization outcomes, quality of life, and patient/caregiver outcomes. The intervention includes comprehensive, standardized palliative care services for adult hepatology cirrhosis patients for which prognosis is poor.

DETAILED DESCRIPTION:
Palliative care is specialized medical care focused on providing patients with relief from the symptoms, pain, and stress of serious or life-limiting illness, regardless of diagnosis, by anticipating, preventing, and treating suffering. Palliative care aims to provide patients and their families with services to help patients make the best possible medical decisions in the face of serious illness. Unfortunately it is often thought to be synonymous with hospice care and therefore underutilized as a part of standard care. Patients with chronic liver disease or cirrhosis may be a particularly underserved population for palliative care, as palliative care may be disregarded until hope of liver transplantation is lost.

Study Description:

* Adult patients admitted to Vanderbilt University Medical Center with cirrhotic advanced liver disease and poor prognosis will be randomized to receive either usual hepatic care or usual hepatic care with comprehensive palliative care services.
* Participants randomized to the intervention arm will receive patient-friendly informational materials, a comprehensive initial palliative care consultation, and follow-up consultations while inpatient. After discharge from hospital, follow-up consults will occur via telephone contact. Telephone contacts will occur on a flexible schedule based on needs and wishes of the participant at a minimum frequency of one contact per month.
* Participants will receive the palliative care intervention for at least 1 year after randomization to the intervention arm or until death.
* Participants randomized to the usual care arm will not be scheduled to meet with the palliative care service unless a meeting is requested by the patient, the family, or treating physician. These consultations include the same palliative care services as the intervention arm, excluding the telephone follow-up consultations.
* All participants will complete quality of life, mood, and satisfaction with care assessments at specified time points for 1 year after randomization or until death. Optional caregiver participation includes completion of satisfaction with care assessments.

Specific aims include:

1. Assess the impact of systematic, comprehensive palliative care services compared to usual hepatic care on time to first hospital readmission within 1-year post randomization.
2. Assess the impact of systematic, comprehensive palliative care services compared to usual hepatic care on other hospital utilization, including days alive out of hospital within 6- months post randomization, total days in hospital (and ICU) within 1-year post randomization, number and cost of hospital admissions within 1-year post randomization, median length of stay per admission, transfers and time to hospice placement, and survival within 1-year post randomization.
3. Assess the impact of systematic, comprehensive palliative care services compared to usual hepatic care on qualify of life.
4. Assess the impact of systematic, comprehensive palliative care services compared to usual hepatic care on patient/caregiver satisfaction.
5. Evaluate the fidelity of the palliative care intervention and assess the generalizability of implementing a large-scale Palliative Care program.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at Vanderbilt University Medical Center with advanced cirrhotic liver disease, whose treating hepatologist indicates a 'No' response to the question, "Would you be surprised if this patient died within 1 year?"

Exclusion Criteria:

* Age < 18 years
* Receipt of liver transplant at the time of potential enrollment
* Inability to give written informed consent (patient or surrogate decision-maker)
* Inability to respond to questions in English
* Treating hepatologist denies permission to enroll
* Receiving hepatology care at non-Vanderbilt sites (to ensure appropriate follow-up)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Bernard, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Started | 31 | 32
Completed | 22 | 20
Not Completed | 9 | 12
Not completed — Death | 9 | 7
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (12.3) | 56.8 (9.4) | 56 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 14 | 18 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 31 | 31 | 62
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 26 | 31 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 63

OUTCOME MEASURES:

1. Primary Outcome: Time to First Hospital Readmission Within 6 Months Post-randomization
Description: Assess the impact of palliative care services on time to first hospital readmission.
  Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: 6 months post-randomization
Population: 5 patients withdrew from the usual hepatic care group and thus only 27 were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 31 | 27
days | 117 [44 to NA] — NA is due to censoring for death and withdrawals. | 68 [22 to NA] — NA is due to censoring for death and withdrawals.

2. Secondary Outcome: Days Alive Out of Hospital
Description: Days alive out of hospital from randomization to 6 months post randomization compared across arms.
  Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: 6 months post-randomization
Population: 5 patients withdrew from the usual hepatic care group and thus only 27 were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 31 | 27
days | 174 [59.5 to 183] | 178 [86.5 to 182.5]

3. Secondary Outcome: Total Days in Hospital
Description: Total days in hospital from randomization to 6 months post randomization compared across arms Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: 6 months post-randomization
Population: 5 patients withdrew from the usual hepatic care group and thus only 27 were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 31 | 27
days | 1 [0 to 10.5] | 3 [0 to 5.5]

4. Secondary Outcome: Total Days in ICU
Description: Total days in ICU from randomization to 6 months post randomization compared across arms.
  Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: 6 months post-randomization
Population: 5 patients withdrew from the usual hepatic care group and thus only 27 were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 31 | 27
Participants
  0 ICU days | 26 | 23
  1 ICU days | 2 | 1
  2 ICU days | 1 | 2
  6 ICU days | 1 | 0
  7 ICU days | 0 | 1
  9 ICU days | 1 | 0

5. Secondary Outcome: Number of Hospital Readmissions
Description: Number of hospital readmissions from randomization to 6 months post randomization compared across arms.
  Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: 6 months post-randomization
Population: 5 patients withdrew from the usual hepatic care group and thus only 27 were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 31 | 27
Participants
  0 readmissions | 15 | 11
  1 readmission | 9 | 8
  2 readmissions | 3 | 5
  3 readmissions | 1 | 2
  4 readmissions | 2 | 1
  5 readmissions | 1 | 0

6. Secondary Outcome: Median Length of Hospital Stay Per Admission
Description: Median length of hospital stay per admission from randomization to 6 months post randomization compared across arms.
  Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: 6 months post-randomization
Population: The sample size indicates number of hospital readmissions per study arm.
Measure: Median (Inter-Quartile Range); unit: days per admission
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 31 | 28
days per admission | 4 [2 to 6] | 2.5 [2 to 5]

7. Secondary Outcome: Hospice Referral
Description: Number of transfers to hospice within 6 months post randomization compared across arms.
  Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: 6 months post-randomization
Population: 5 patients withdrew from the usual hepatic care group and thus only 27 were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 31 | 27
Participants | 1 | 4

8. Secondary Outcome: Time to Hospice Placement
Description: Number of days from hospice referral to time to hospice placement. Time frame was changed from 1 year to 6 months due to early termination. There are only 3 patients with a hospice admission date that is after baseline discharge, all of whom are from the control group. The remaining patients with hospice referral but are missing a hospice admission date due to death before hospice admission. Therefore, it is not feasible to calculate any statistics.
Time Frame: 6 months post-randomization
Population: There are only 3 patients with a hospice admission date that is after baseline discharge, all of whom are from the control group. The remaining patients with hospice referral but are missing a hospice admission date due to death before hospice admission. Therefore, it is not feasible to calculate any statistics.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 0 | 3
Participants
  4.36 days |  | 1
  2.78 days |  | 1
  143.84 days |  | 1

9. Secondary Outcome: Change in Chronic Liver Disease Questionnaire (CLDQ)
Description: Change in liver disease-related quality of life: The CLDQ is a 29-item questionnaire measuring 6 domains. Item scores range from 1 to 7 with higher scores indicating better quality of life. The total score can range from 29 to 203 with a score of 1 meaning the symptom being assessed is "present always" while a score of 7 means the symptom is "never present". Therefore, a higher score corresponds to a better quality of life while a lower score corresponds to a worse quality of life. The questions in each domain have a range of factor loads indicative of their impact, and a clinically important difference is defined as a score change of 0.5.
  Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: Change from baseline over 6 months post-randomization
Population: Only 5 participants in each group returned both the baseline and 6-month surveys.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 5 | 5
score on a scale | 0.52 [0.34 to 1.41] | 0.34 [-0.1 to 0.7]

10. Secondary Outcome: Change in EQ-5D-5L
Description: Change in generic health status: The EQ-5D-5L is a 5-item questionnaire with responses ranging from absence of symptom to extreme experience of the symptom. This scale is numbered from 0 to 100. 100 means the best health you can imagine and 0 means the worst health you can imagine.
  Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: Change from baseline over 6 months post-randomization
Population: Only 5 participants from each group returned both baseline and 6-month surveys.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 5 | 5
score on a scale | 21 [-5 to 31] | -1 [-7 to 20]

11. Secondary Outcome: Change in PROMIS Emotional Distress - Anxiety - Short Form 4a
Description: Change in mood (anxiety): The PROMIS Emotional Distress - Anxiety - Short Form 4a contains 4 items that measure anxiety on a 5-point Likert scale with higher scores indicating increased symptomatology. The raw score can range from 4 to 20 which converts to a t-score range of 40.3 to 81.6.
  Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: Change from baseline over 6 months post-randomization
Population: Only 5 participants from each group returned both baseline and 6-month surveys.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 5 | 5
score on a scale | 0 [-1 to 0] | 0 [0 to 2]

12. Secondary Outcome: Change in PROMIS Emotional Distress - Depression - Short Form 4a
Description: Change in mood (depression): The PROMIS Emotional Distress - Depression - Short Form 4a contains 4 items that measure depression on a 5-point Likert scale with higher scores indicating increased symptomatology. The raw score ranges from 4 to 20 which converts to a t-score range of 41.0 to 79.4.
  Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: Change from baseline over 6 months post-randomization
Population: Only 4 participants from the comprehensive palliative care services each group and 5 participants from the usual hepatic care group returned both baseline and 6-month surveys.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 4 | 5
score on a scale | -4 [-7.95 to -2.17] | -3.2 [-3.5 to 1.9]

13. Secondary Outcome: Change in Satisfaction With Care (Quality of End-of-Life Care: Questionnaire for Patient)
Description: Change in patient satisfaction with care: The Quality of End-of-Life Care: Questionnaire for Patient is an 11-item questionnaire, with items scored on a 10-point Likert type scale with higher scores indicating better satisfaction with care. The score can range from 0 to 110.
  Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: Change from baseline over 6 months post-randomization
Population: Only 5 participants from the comprehensive palliative care services each group and 4 participants from the usual hepatic care group returned both baseline and 6-month surveys.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 5 | 4
score on a scale | 0 [0 to 3.25] | 0.8 [-0.91 to 1.96]

14. Secondary Outcome: Change in Kingston Caregiver Stress Scale
Description: The Kingston Caregiver Stress Scale will be used to measure caregiver stress. The KCSS is designed to measure stress experienced by lay caregivers, not institutional staff, and was designed to monitor change in an individuals stress over time. Ten items are grouped into three categories: care giving, family, and financial issues. Scores can range from 10 to 50. Lower scores indicate less stress and higher scores indicate high stress.
  Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: Change from baseline over 6 months post-randomization
Population: The intended population included caregivers. There is no statistics to report. The two scores from participants in the intervention group are indicated below.
Measure: Count of Participants; unit: Participants
Groups:
- Comprehensive Palliative Care Services - Caregivers: Comprehensive Palliative Care services in addition to usual hepatic care
  Comprehensive Palliative Care services: Participants who are randomly assigned to the intervention arm will receive informational materials, comprehensive inpatient palliative care consultations with a palliative care physician or nurse practitioner, in addition to standard hepatic care. If the patient is discharged, follow-up consults will be provided by a palliative care nurse via telephone contact. Telephone contacts will occur on a flexible schedule (e.g., weekly, bi-weekly, monthly) based on the needs and wishes of the patient, at a minimum frequency of once a month. If a need for further care is identified from a telephone contact, appropriate follow-up (referral, appointment, clinical communication, etc.) will occur per standard procedures. If the participant is readmitted, the consultation schedule will restart.
- Usual Hepatic Care - Caregivers: Usual hepatic care
  Usual hepatic care: Participants randomized to the usual care arm will not be scheduled to meet with the palliative care service unless a consult is requested by the patient, the family, or treating physician. These consultations would include the same palliative care services as the intervention arm, excluding the informational patient materials and telephone consultations.
Arm/Group | Comprehensive Palliative Care Services - Caregivers | Usual Hepatic Care - Caregivers
Number analyzed (Participants) | 2 | 0
Participants
  Change in Kingston Caregiver Stress Scale Score:15 | 1 |
  Change in Kingston Caregiver Stress Scale Score:7 | 1 |

15. Secondary Outcome: Change in Satisfaction With Care (Quality of End-of-Life Care: Questionnaire for Patient Adapted for Caregiver)
Description: Change in caregiver satisfaction with care: The Quality of End-of-Life Care: Questionnaire for Patient item wording was modified to apply to caregivers. The questionnaire is an 11-item questionnaire, with items scored on a 10-point Likert type scale with higher scores indicating better quality of care. The score can range from 0 to 110.
  Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: Change from baseline over 6 months post-randomization
Population: The intended population includes the caregivers. Only one caregiver in each group returned both surveys.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Comprehensive Palliative Care Service - Caregivers: Comprehensive Palliative Care services in addition to usual hepatic care
  Comprehensive Palliative Care services: Participants who are randomly assigned to the intervention arm will receive informational materials, comprehensive inpatient palliative care consultations with a palliative care physician or nurse practitioner, in addition to standard hepatic care. If the patient is discharged, follow-up consults will be provided by a palliative care nurse via telephone contact. Telephone contacts will occur on a flexible schedule (e.g., weekly, bi-weekly, monthly) based on the needs and wishes of the patient, at a minimum frequency of once a month. If a need for further care is identified from a telephone contact, appropriate follow-up (referral, appointment, clinical communication, etc.) will occur per standard procedures. If the participant is readmitted, the consultation schedule will restart.
Arm/Group | Comprehensive Palliative Care Service - Caregivers | Usual Hepatic Care - Caregivers
Number analyzed (Participants) | 1 | 1
score on a scale | 0 [0 to 0] | -2.83 [-2.83 to -2.83]

16. Secondary Outcome: Liver Transplant Status
Description: Number of deferred, listed, and declined listing for liver transplant compared across arms.
  Time frame was changed from 1 year to 6 months due to early termination. Liver transplant status data was not obtained.
Time Frame: 6 months post-randomization
Population: Liver transplant status data was not obtained.
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Model for End-Stage Liver Disease (MELD) Score
Description: Baseline MELD score compared across arms. MELD score ranks the participants degree of sickness and indicates how much the participant needs a liver transplant. The score ranges from 6-40. The higher the number the more urgent the need for a transplant.
Time Frame: Baseline
Population: Baseline MELD scores were only available for 26 intervention group participants and 27 control group participants.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 26 | 27
score on a scale | 24 [20 to 26] | 24 [17.5 to 28]

18. Secondary Outcome: Completed Liver Transplants
Description: Number of patients with completed liver transplants compared across arms. Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: 6 months post-randomization
Population: 5 participants withdrew from the usual hepatic care group.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 31 | 27
Participants | 4 | 3

19. Secondary Outcome: Physical Symptoms
Description: Number of documented physical symptoms (ascites, variceal bleeding, encephalopathy, etc.) compared across arms.
  Time frame was changed from 1 year to 6 months due to early termination. Physical symptom data was not obtained.
Time Frame: 6 months post-randomization
Population: Physical symptom data was not obtained.
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Presence of Advance Directives
Description: Percentage of patients with documented advance care directives compared across arms.
  Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: 6 months post-randomization
Population: 5 participants withdrew from the usual hepatic care group.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 31 | 27
Participants | 25 | 23

21. Secondary Outcome: Survival
Description: Survival rate compared across arms. Time frame was changed from 1 year to 6 months due to early termination.
Time Frame: 6 months post-randomization
Population: 5 participants withdrew from the usual hepatic care group.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
Number analyzed (Participants) | 31 | 27
Participants | 22 | 20

22. Secondary Outcome: Provider Satisfaction
Description: The "ICU Provider Satisfaction Survey with the Palliative Care Program:Veterans Affairs of Ann Arbor" instrument is available online and has been modified for the current study by removing the 'ICU' reference and revising 'pain' to symptoms more relevant to the current population. The survey includes 7-item questionnaire, with items scored on a 5-point Likert type scale with higher scores indicating better provider satisfaction. The score can range from 0 to 35.
  Time frame was changed due to early termination. Data was not collected.
Time Frame: Change from Baseline to study closeout.
Population: The provider population was not analyzed because data was not collected.
Groups:
- Comprehensive Palliative Care Services - Providers: Comprehensive Palliative Care services in addition to usual hepatic care
  Comprehensive Palliative Care services: Participants who are randomly assigned to the intervention arm will receive informational materials, comprehensive inpatient palliative care consultations with a palliative care physician or nurse practitioner, in addition to standard hepatic care. If the patient is discharged, follow-up consults will be provided by a palliative care nurse via telephone contact. Telephone contacts will occur on a flexible schedule (e.g., weekly, bi-weekly, monthly) based on the needs and wishes of the patient, at a minimum frequency of once a month. If a need for further care is identified from a telephone contact, appropriate follow-up (referral, appointment, clinical communication, etc.) will occur per standard procedures. If the participant is readmitted, the consultation schedule will restart.
- Usual Hepatic Care - Providers: Usual hepatic care
  Usual hepatic care: Participants randomized to the usual care arm will not be scheduled to meet with the palliative care service unless a consult is requested by the patient, the family, or treating physician. These consultations would include the same palliative care services as the intervention arm, excluding the informational patient materials and telephone consultations.
Arm/Group | Comprehensive Palliative Care Services - Providers | Usual Hepatic Care - Providers
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: baseline to 6 months
Arm/Group | Comprehensive Palliative Care Services | Usual Hepatic Care
All-Cause Mortality (participants affected / at risk) | 9/31 | 7/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 0/31 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT03022630/Prot_SAP_000.pdf